CLINICAL TRIAL: NCT01529229
Title: A Double-blind, Randomized, Multicenter Parallel-group Study on Efficacy of Desloratadine and Prednisolone Association Compared to Dexchlorpheniramine and Betamethasone Association in Children (2-12 Years) With Moderate - Severe Persistent Allergic Rhinitis
Brief Title: Comparison of Desloratadine Associated With Prednisolone Oral Solution Versus Dexchlorpheniramine Associated With Betamethasone for Persistent Allergic Rhinitis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPREMS1111
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — dexchlorpheniramine; Betamethasone; desloratadine; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desloratadine + Prednisolone (Experimental): Desloratadine(0.5 mg/ml) Associated With Prednisolone (4 mg/ml) Oral Solution once a day - bottle 1 + placebo 2 times a day - bottles 2 and 3.
  Interventions: Drug: Desloratadine + Prednisolone
- Dexchlorpheniramine + Betamethasone (Active Comparator): Dexchlorpheniramine (0.4 mg/ml) + Betamethasone (0.05 mg/ml) three times a day - bottles 1, 2 and 3.
  Interventions: Drug: Dexchlorpheniramine + Betamethasone

INTERVENTIONS:
Drug: Dexchlorpheniramine + Betamethasone — Children (2 to 5 years): 2.5 ml 3 times a day Children (6 to 12 years): 5.0 ml 3 times a day
  Arms: Dexchlorpheniramine + Betamethasone
Drug: Desloratadine + Prednisolone — Children (2 to 5 years): 2.5 ml 3 times a day Children (6 to 12 years): 5.0 ml 3 times a day
  Arms: Desloratadine + Prednisolone

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drug associations in the treatment of Moderate - Severe Persistent Allergic Rhinitis.

DETAILED DESCRIPTION:
* double-blind, non-inferiority, prospective, parallel group trial.
* Experiment duration: 07 days.
* 02 visits (days 0 and 7).
* Efficacy will be evaluated for persistent allergic rhinitis based on nasal symptoms score
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the patient or legal guardian;
* Clinical diagnosis of moderate - severe persistent allergic rhinitis according to the classification of ARIA (Allergic Rhinitis and Its Impact on Asthma);
* Children aged between 2 and 11 years and 11 months (up to 30 kg);
* Presence of nasal symptoms score greater than or equal to 5 (scale 0 to 12)in the last week;
* Evidence of sensitization to aeroallergens in examination (immediate skin tests or serum specific IgE) in the 12 months prior to inclusion.

Exclusion Criteria:

* Participation in clinical trial in 30 days prior to study entry;
* Patients receiving immunotherapy;
* Patients with history of hypersensitivity to desloratadine or prednisolone or with corticosteroids use contraindications ;
* Patients with any clinically significant disease other than allergic rhinitis, including hematopoietic, cardiovascular, renal, neurological, psychiatric or autoimmune disorders;
* Patients on treatment with monoamine oxidase inhibitors (MAOIs);
* Patients who were in use of oral antihistamines or decongestants in the past 15 days;
* Patients who were treated with systemic corticosteroids in the last month;
* Patients who have uncontrolled asthma, chronic sinusitis, drug related rhinitis and nasal anatomic abnormalities.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in persistent allergic rhinitis based on nasal symptoms score | 7 days
  The mean variability of nasal symptoms score observed between visit 1 and visit 2 will be used as the primary endpoint of clinical efficacy.

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 7 days
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Solé, MD, Principal Investigator — Federal University of São Paulo